CLINICAL TRIAL: NCT05428462
Title: Effectiveness of a One-day Psychoeducation Program on Internalized Stigmatization for Borderline Personality Disorder (BPD) Patients
Brief Title: Effectiveness of a One-day Psychoeducation Program on Internalized Stigmatization for BPD Patients
Acronym: EDUC-BPD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0611
Record Dates: First submitted 2022-06-16; First posted 2022-06-23 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-05

CONDITIONS: Borderline Personality Disorder
Keywords: Psychoeducation day; internalized stigmatization
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Psychoeducation day on borderline personality disorder — Transmission of latest knowledge on borderline personality disorder

SUMMARY:
Education day on borderline personality disorder (BPD), including a transmission of current scientific knowledge on the disease. A dimensional understanding of BPD is delivered as well as disidentification of oneself to the symptoms of borderline personality disorder (Ducasse 2020 Eur Arch Psychiatry Clin Neurosci). The main objective is to evaluate the impact of borderline education day on self-stigma.

DETAILED DESCRIPTION:
Borderline personality disorder defined as "a pattern of instability in interpersonal relationships, self-image and affects, and impulsiveness marked" concerns 4-6% of the general population. This is the emotional trouble the most associated with the occurence of suicide attempts (85% of these patients make multiple suicide attempts) and death by suicide (10% of these patients). This is a major public health problem.

A large number of patients with borderline personality disorder are not informed of their diagnosis. The main reasons are : the non-recognition of this disorder by health professionals, the belief that borderline personality disorder is a overly stigmatizing diagnosis , or preference to diagnose another disorder - that professionals think respond better to treatments and therefore be of a better prognosis.

Patients with borderline personality disorder often think themselves as "bad people" or the only people suffering from these symptoms. Thus, the ignorance of borderline personality disorder by patients leads to a basis of their altered sense of identity, perceived as defective or isolated. This generate a strong internalized stigma.

Many people diagnosed with borderline personality disorder receive no information about this disorder while psychoeducation has shown its effectiveness in severe psychiatric disorders, including the disorder of borderline personality, by reducing the negative repercussions psychiatric pathology. Moreover, the education of patients suffering from self-stigma makes it possible to in the face of negative beliefs around the disease and the acquisition of knowledge about the disorder and how to deal with it reduces self-stigma in bipolar patients. However, the propensity to feel shame - the stigmatization of oneself as worthless - is strongest in borderline personality disorder compared to all psychiatric disorders and most associated with the occurence of suicidal behaviors. In recommendations with good clinical practice, the investigator propose within the sector a day of education on borderline personality disorder including a transmission of current scientific knowledge on the illness, a dimensional understanding of the disorder, and the dis-identification of self to the symptoms of borderline personality disorder. The investigator hypothesize that this day of psychoeducation makes it possible to decrease self-stigma, which could be a mediator in reducing negative repercussions of borderline pathology.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Borderline Personality disorder assessed according to SCID II
* Having attended the borderline education day

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is patients with Borderline Personality disorder assesed according to the SCID II
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of internalized stigma of mental illnessillness | At immediate post-intervention
  Comparison of internalized stigma of mental illness between pre-treatment
Comparison of internalized stigma of mentalillness | At 3 months post-intervention
  Comparison of internalized stigma of mental illness between pre-treatment

SECONDARY OUTCOMES:
Depressive symptoms using the Beck Depression Inventory | At immediate post-intervention
  Comparison of depressive symptoms between pre-treatment and post-intervention
Depressive symptoms using the Beck Depression Inventory | At 3 months post-intervention
  Comparison of depressive symptoms between pre-treatment and 3 months post-intervention
Severity of suicidal ideation evaluated by the likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At immediate post-intervention
  Comparison of the intensity of suicidal ideation between pre-treatment and post-intervention
Severity of suicidal ideation evaluated by the likert scales from 0 (none) to 10 (maximum possible suicidal ideation) | At 3 months post-intervention
  Comparison of the intensity of suicidal ideation between pre-treatment and 3 months post-intervention
Psychological pain using the Likert scales from 0 (none) to 10 (maximum possible pain) | At immediate post-intervention
  Comparison of psychological pain between pre-treatment and post-intervention
Psychological pain using the Likert scales from 0 (none) to 10 (maximum possible pain) | At 3 months post-intervention
  Comparison of psychological pain between pre-treatment and 3 months post-intervention
The intensity of hopelessness using the Likert scales from 0 (none) to 10 (maximum possible hopelessness) | At immediate post-intervention
  Comparison of the intensity of hopelessness between pre-treatment and post-intervention
The intensity of hopelessness using the Likert scales from 0 (none) to 10 (maximum possible hopelessness) | At 3 months post-intervention
  Comparison of the intensity of hopelessness between pre-treatment and 3 months post-intervention
The intensity of optimism using analog visual scale | At immediate post-intervention
  Comparison of the intensity of optimism between pre-treatment and post-intervention
The intensity of optimism using analog visual scale | At 3 months post-intervention
  Comparison of the intensity of optimism between pre-treatment and 3 months post-intervention
Feeling of pleasure using the quality of life questionnaire on pleasure and satisfaction | At immediate post-intervention
  Comparison of feeling of pleasure between pre-treatment and post-intervention
Feeling of pleasure using the quality of life questionnaire on pleasure and satisfaction | At 3 months post-intervention
  Comparison of feeling of pleasure between pre-treatment and 3 months post-intervention
Feeling of satisfaction using the quality of life questionnaire on pleasure and satisfaction | At immediate post-intervention
  Comparison of feeling of satisfaction between pre-treatment and post-intervention
Feeling of satisfaction using the quality of life questionnaire on pleasure and satisfaction | At 3 months post-intervention
  Comparison of feeling of satisfaction between pre-treatment and 3 months post-intervention
Anxiety state using the State-Trait Inventory (STAI-State) | At immediate post-intervention
  Comparison of the state of anxiety between pre-treatment and post-intervention
Anxiety state using the State-Trait Inventory (STAI-State) | At 3 months post-intervention
  Comparison of the state of anxiety between pre-treatment and 3 months post-intervention
Hopelessness using the Beck Hopelessness Scale (BHS) | At immediate post-intervention
  Comparison of the hopelessness between pre-treatment and post-intervention
Hopelessness using the Beck Hopelessness Scale (BHS) | At 3 months post-intervention
  Comparison of the hopelessness between pre-treatment and 3 months post-intervention
Level of positive and negative affects using the PANAS Scale | At immediate post-intervention
  Comparison of level of positive and negative affects between pre-treatment and post-intervention
Level of positive and negative affects using the PANAS Scale | At 3 months post-intervention
  Comparison of level of positive and negative affects between pre-treatment and 3 months post-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC